CLINICAL TRIAL: NCT05949736
Title: Effect of Telemedicine Music Therapy in Medical Students With Depression, Anxiety, or Insomnia.
Brief Title: Effect of Music Therapy in Medical Students (EMTMS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Province Nanjing Brain Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 81725005-6
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Depression; Anxiety; Insomnia
Keywords: Telemedicine; Music Therapy; Mental sub-health; Acoustic features; Wearable devices; Functional near-infrared evaluation
MeSH Terms: conditions — Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Clinical Symptom Changes of Music Therapy in a Randomized Controlled Study. (Experimental): This study investigates the clinical symptom changes of the Music Therapy (MT) group through a randomized controlled trial, aiming to explore the short- and long-term efficacy of MT for individuals experiencing mental sub-health. The study includes one-month and six-month post-treatment follow-ups to assess the lasting effects of MT intervention.
  Interventions: Device: The Online intervention platform
- The changes of objective markers of the music therapy. (Experimental): This study examines the changes in objective markers resulting from Music Therapy (MT) intervention. It explores alterations in behavior, biological features, and neuroimaging data to understand the potential biological mechanism underlying the efficacy of music therapy. By analyzing these objective markers, the study aims to gain valuable insights into the impact of MT on individuals' mental well-being.
  Interventions: Device: The Online intervention platform

INTERVENTIONS:
Device: The Online intervention platform — Music Therapy (MT) is known to have a calming effect on individuals by using relaxing and soothing music, gradually inducing a state of relaxation. Moreover, it can effectively regulate individual psychological emotions through its influence on specific brain regions such as the cerebral cortex, hypothalamus, and limbic system. This regulation of emotional responses can lead to an improvement in daily mood, reducing feelings of tension and anxiety.

SUMMARY:
Mental health has become an increasingly pressing concern, especially since the onset of the COVID-19 pandemic. However, not all individuals experiencing mental suboptimal states require pharmacological treatment. Telemedicine offers psychological interventions like Music Therapy (MT), which utilizes remote network technology to provide effective psychological services. MT achieves its therapeutic effect by improving the brain's internal network activation patterns, thus promoting self-regulation. With relaxing and soothing music, MT gradually helps individuals unwind and regulates their psychological emotions by influencing the cerebral cortex, hypothalamus, and limbic system, leading to an improved daily mood and reduced tension and anxiety.

The study was designed as a randomized clinical trial, comprising a telemedicine intervention group (MT) and a waiting control group (CON group), both of whom were in a state of mental sub-health. The MT group received music therapy, while the Waiting group received the MT intervention after the treatment of the MT group.

The aim of this study was to collect mental health symptom data, behavioral data, and voice expression data using mobile phone, wearable devices (WD) and neuroimaging techniques (fNIRS). These indicators were used as objective measures to assess the long-term and short-term efficacy of telep-sychological interventions. Analyzing digital biomarkers allowed for a deeper understanding of the potential biological and neurobiological mechanisms underlying the effectiveness of tele-psychological interventions.

DETAILED DESCRIPTION:
The Internet intervention study is a double-blind randomized controlled trial designed to assess the efficacy of Internet-based Music Therapy (MT) compared to a waiting control group for individuals experiencing mental sub-health. Participants will be randomly assigned in a 1:1 ratio to either the intervention group (MT group) or the waiting group (CON group).

Participants in the MT group will receive 12 sessions, spread over a 3-4 week period, with 3-4 sessions per week, each lasting 20-30 minutes. The MT group will undergo music therapy during the first 4 weeks. Clinical symptom assessments and related data will be collected from participants before MT (baseline) and after MT (at the 3rd or 4th week, 1 month, and 6 months). The MT sessions will be divided into three stages, each focusing on a specific topic: Physical and mental relaxation stage: Participants will learn relaxation techniques encompassing the whole body and mind, including breathing and muscle relaxation. Nature imagination stage: Guided music imagination will be utilized during this stage. Internal self-exploration: Participants will explore positive experiences and potential within themselves, adopting a resource-oriented approach for psychological intervention. Participants in the CON group will not receive any intervention during the treatment of the MT group.

Throughout the study, all participants will undergo symptom assessment, poetry reading, voice collection, functional near-infrared evaluation (fNIRS), and wearable devices monitoring to collect data.

The study aims to achieve the following objectives: Evaluate changes in clinical symptoms, such as depression, anxiety, or insomnia, after the telemedicine MT intervention for individuals experiencing mental sub-health. Gain deeper insights into the possible biological mechanisms underlying the efficacy of tele-MT intervention by analyzing digital biomarkers. Explore the predictive effect of objective biomarkers on the treatment outcomes of tele-MT. The study's ultimate goal is to contribute to the understanding and effectiveness of telemedicine-based MT interventions for individuals facing mental sub-health.

ELIGIBILITY:
Inclusion Criteria:

Participants with a total score of PHQ-9 >5 or a total score of GAD-7 >5 or a total score of ISI >7 will be eligible to participate in the study.

Exclusion Criteria:

1. Participants with self-reported lifetime suicide attempt, active self-harm, or active suicidal ideation with intent will be excluded from the study.
2. Participants with a clinician-diagnosed bipolar disorder, substance use disorder, or any psychotic disorder, including schizophrenia, will not be eligible to participate.
3. Individuals who are incapable of understanding or completing study procedures and digital intervention, as determined by the participant, patient/legal guardian, healthcare provider, or clinical research team, will be excluded.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in depressive symptoms assessed by the Patient Health Questionnaire-9 (PHQ-9; range: 0-27) at week 4, week 8, and week 28. | Baseline, 4th week, 8th week, and 28th week.
  The total scores of these questionnaires were interpreted as follows: normal (0-4), mild (5-9), moderate (10-14), and severe (15-27) depression.
Change from baseline in anxiety symptoms assessed by the Generalized Anxiety Disorder-7 (GAD-7, range: 0-21) at week 4, week 8, and week 28. | Baseline, 4th week, 8th week, and 28th week.
  TThe total scores of these questionnaires were interpreted as follows: normal (0-4), mild (5-9), moderate (10-14), and severe (15-21) anxiety.
Change from baseline in insomnia symptoms assessed by the Insomnia Severity Index (ISI; range: 0-28) at week 4, week 8, and week 28. | Baseline, 4th week, 8th week, and 28th week.
  The total scores of these questionnaires were interpreted as follows: normal (0-7), mild (8-14), moderate (15-21), and severe (22-28) insomnia.

SECONDARY OUTCOMES:
Change from baseline in perceived stress assessed by the Perceived Stress Scale-14 (PSS-14; range: 0-56) at week 4, week 8, and week 28. | Baseline, 4th week, 8th week, and 28th week.
  The total scores of these questionnaires were interpreted as follows: normal (0-28), moderate (29-42), severe (43-56).
Change from baseline in suicidal ideation assessed by the Beck Scale for Suicide (BSS-14; range: 0-38) at week 4, week 8, and week 28. | Baseline, 4th week, 8th week, and 28th week.
  The total scores of these questionnaires were interpreted as follows: no or low suicidal ideation (0-8), moderate suicidal ideation (9-16), high suicidal ideation (17-38).
Change from baseline in behavioral data measured by wearable devices (WD) during treatment. | Baseline to 4th week.
  The behavioral data include heart rate (bpm), blood oxygen (SaO2), sleep time (s), and the number of steps.
Change from baseline in acoustic features. | Baseline, 4th week, 8th week, and 28th week.
  Participants will record videos prior to beginning intervention (baseline) and after completing intervention (week 4, week 8, and week 28). Acoustic features (Hz) are a set of indicators that can reflect an individual's emotional state.
The neuro-changes resulting from the MT intervention. | Baseline, 2th week, and 4th week.
  The functional near-infrared spectroscopy (fNIRS) data will be collected at three time points: before MT intervention, at the end of intervention section 6, and after the entire intervention treatment. The fNIRS can collect the oxygenated hemoglobin and deoxyhemoglobin during brain activity.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Wang, Ph.D, Study Chair — Affiliated Nanjing Brain Hospital, Nanjing Medical University
Locations (3):
- China (3):
  - Hainan Medical College, Haikou, Hainan
  - Xinxiang Medical University, Xinxiang, Henan
  - Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No